CLINICAL TRIAL: NCT07314151
Title: Study on the Use of Traditional Chinese Medicine Diagnostic Tools to Assist in Identifying the Clinical Characteristics of Inflammatory Bowel Disease and Research on Metabolic Plastids of Tongue Coating
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH113-REC2-014
Record Dates: First submitted 2025-12-08; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis)
Keywords: inflammatory bowel disease, Crohn's disease, ulcerative colitis, gut brain axis, Traditional Chinese medicine (TCM) diagnosis, Tongue diagnosis, Metabolomics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD Patient Cohort
  Interventions: Other: No intervention (observational study with diagnostic assessments only)
- Healthy Control Cohort
  Interventions: Other: No intervention (observational study with diagnostic assessments only)

INTERVENTIONS:
Other: No intervention (observational study with diagnostic assessments only) — This observational study involves no therapeutic or behavioral intervention. Participants undergo non-invasive assessments including Traditional Chinese Medicine four-diagnostic measurements (inspection, listening/smelling, inquiry, and pulse assessment), completion of standardized questionnaires, and collection of tongue-coating samples for metabolomic analysis.

SUMMARY:
This study will be conducted at the outpatient clinic of China Medical University hospital. It is expected to enroll two groups of 30 subjects, including the experimental group must meet the clinical diagnosis of IBD, and the control group without IBD and have no obvious gastrointestinal symptoms . This proje ct uses modern TCM diagnostic tools, such as tongue diagnosis instrument, auscul tation instrument, TCM constitution questionnaire, and pulse diagnosis instrument to establish the comparison of physiological and biochemical indicators such as TCM phenotype and laboratory tests data in patients with IBD. Besides, another purpose of this project is to analyze the tongue coating metabolites of patients with IBD by mass spectrometry, and to establish a research model of tongue coating an d metabolomics for patien ts with IBD and the prognosis analysis of acute and remission phases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older who are able to provide informed consent and comply with the study procedures.
* Experimental group: Patients with a primary diagnosis of Crohn's disease or ulcerative colitis, defined by ICD-10-CM codes K50-K51.
* Control group: Individuals without inflammatory bowel disease and without significant gastrointestinal symptoms.

Exclusion Criteria:

* Individuals who are unable to provide informed consent or unable to comply with study procedures or questionnaires.
* Individuals who have undergone major surgery or received chemotherapy or radiotherapy within the past month.
* Pregnant women.
* Individuals deemed unsuitable for participation in this study by the attending physician.
* Control group exclusions:

  * Individuals with any diagnosed psychiatric disorder.
  * Individuals with any major gastrointestinal disease, such as gastrointestinal malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the outpatient clinics of China Medical University Hospital and is designed to enroll two groups of participants, with 100 individuals aged 18 years or older in each group. The experimental group will include patients who meet the clinical diagnostic criteria for inflammatory bowel disease (IBD), while the control group will consist of individuals without IBD and without significant gastrointestinal symptoms.
  All participants will receive a detailed explanation of the study from research personnel. Those who agree to participate and pass the initial screening will be required to sign an informed consent form for human clinical research and subsequently undergo the relevant assessments and procedures.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Tongue-coating metabolomic profiles in patients with inflammatory bowel disease compared with healthy controls | At enrollment (single visit; cross-sectional assessment)
  After tongue-coating collection, the samples (approximately 20-50 mg) are weighed and stored at -80 °C until all samples have been collected. Metabolite extraction is then performed, followed by analysis of metabolite signals using liquid chromatography-mass spectrometry. The primary analytical platform consists of an ACQUITY UPLC I-Class System (Waters) coupled with a Vion IMS Q-ToF mass spectrometer (Waters).
  The acquired chromatographic and mass spectrometric data are further processed using the omics analysis software Progenesis QI to identify intergroup differences. Metabolite signal differences between the acute and remission phases are evaluated using principal component analysis (PCA) and partial least squares discriminant analysis (PLS-DA). Subsequently, differential metabolite signals are matched against reference databases for metabolite identification. Upon completion of metabolite identification and data acquisition, disease phase-specific metabolomic signature patterns

SECONDARY OUTCOMES:
Constitution in Chinese Medici n e Questionnaire, CCMQ | At enrollment (single visit; cross-sectional assessment)
  During participant enrollment, questionnaires are administered by research personnel. Participants are instructed to complete the questionnaires independently based on their subjective perceptions, with efforts made to minimize external interference that may influence their responses. Questionnaire results are scored and categorized according to the established scoring criteria.
Gastrointestinal Symptom Rating Scale , GSRS | At enrollment (single visit; cross-sectional assessment)
  The Gastrointestinal Symptom Rating Scale (GSRS) assesses 15 common gastrointestinal symptoms grouped into five symptom domains: abdominal pain, diarrhea, gastroesophageal reflux, indigestion, and constipation. Each item is rated on a 7-point Likert scale ranging from "no discomfort" to "very severe discomfort," with participants self-assessing the severity of their gastrointestinal symptoms over the preceding week. Higher scores indicate greater symptom severity.
  The GSRS provides a brief yet comprehensive assessment of common gastrointestinal symptoms and demonstrates good internal consistency and psychometric validity. The reported Cronbach's alpha values range from 0.74 to 0.85, and the test-retest reliability ranges from 0.55 to 0.70.
Hospital Anxiety and Depressio n Scale, HADS | At enrollment (single visit; cross-sectional assessment)
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items, with 7 items assessing anxiety (HADS-A) and 7 items assessing depression (HADS-D), each scored separately. Items are rated on a 4-point scale ranging from 0 to 3, with higher scores indicating greater severity of anxiety or depression. According to the original authors' recommendations, scores of 7 or below indicate no anxiety or depression, scores of 8-10 suggest possible anxiety or depression, and scores of 11 or higher indicate a high likelihood of clinically significant anxiety or depression.
Crohn's Disease Activity Index CDAI | At enrollment (single visit; cross-sectional assessment)
  The assessment consists of eight clinical variables, including subjective symptoms over the preceding week (such as abdominal pain severity and overall well-being), objective measures (such as the use of antidiarrheal medications and percentage change in body weight), and laboratory parameters. After individual component scores are recorded, a weighted calculation is applied to generate the total score. Higher scores indicate greater disease activity, with a CDAI score of less than 150 indicating disease remission and a score greater than 450 indicating extremely severe disease activity.
Partial Mayo Scoring Index, pM ayo | At enrollment (single visit; cross-sectional assessment)
  The partial Mayo (pMayo) scoring index primarily records stool frequency, rectal bleeding, and physician's global assessment in patients with ulcerative colitis. Each component is scored on a scale of 0 to 3, yielding a total score ranging from 0 to 9, with higher scores indicating greater disease activity. The pMayo score demonstrates a specificity of 0.84 for identifying disease remission and a sensitivity of 0.71.
Tongue diagnostic device | At enrollment (single visit; cross-sectional assessment)
  Tongue images are captured from a frontal view with the participant's head stabilized on the tongue diagnostic examination platform. Each participant is instructed to protrude the tongue naturally during image acquisition. After image capture, the images are transmitted to a computer for processing. The photographs are first calibrated using a standard color reference card to correct pixel color deviations, and tongue features are subsequently analyzed using a computer-assisted interpretation system to support Traditional Chinese Medicine tongue diagnosis. The assessed tongue features include:
  1. Tongue shape: small, medium, or enlarged.
  2. Tongue color: pale, light red, red, or purplish.
  3. Tongue body features: red dots, petechiae/ecchymosis, teeth marks, and fissures.
  4. Coating color: white or yellow.
  5. Coating thickness: scant, thin, or thick.
  6. Saliva (moisture): scant, normal, or excessive.
  7. Sublingual collateral veins: normal or abnormal.
Listening diagnostic device | At enrollment (single visit; cross-sectional assessment)
  The listening diagnostic device is based on a computerized acoustic analysis system that provides functions for voice signal analysis and management of participants' voice data. The core technology involves recording a one-second sustained vowel sound (e.g., /a/) to quantify acoustic parameters and perform model-based analyses. Medical research and published studies have demonstrated that the derived parameters are capable of distinguishing deficiency-related constitutional characteristics among different participants, making this system a practical diagnostic tool for rapid constitutional assessment during Traditional Chinese Medicine clinical syndrome differentiation.
Pulse diagnostic device | At enrollment (single visit; cross-sectional assessment)
  Clinical pulse signals are analyzed using time-domain methods to evaluate pulse position, rate, rhythm, and waveform characteristics The system automatically interprets Traditional Chinese Medicine syndrome patterns to assist physicians in clinical diagnosis and syndrome differentiation.
  Using the pulse diagnostic device, objective and quantifiable parameters can be obtained, including pulse waveform data, blood pressure (systolic/diastolic), heart rate (beats per minute), cardiac arrhythmia indices (number of irregular heartbeats within a five-minute period), heart rate variability (HRV; overall autonomic nervous system activity), low-frequency power (LF; sympathetic nervous system activity), high-frequency power (HF; parasympathetic nervous system activity), and the LF/HF ratio, which reflects the balance between sympathetic and parasympathetic nervous system activity.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North, Taiwan